CLINICAL TRIAL: NCT00742794
Title: Frequency of Hymenoptera-stings in Patients Under and After Allergen-specific Immunotherapy: a Retrospective Data-analysis Considering Socio-economic Aspects
Brief Title: Frequency of Hymenoptera-stings in Patients Under Allergen-Specific Immunotherapy (SIT)
Acronym: ZU-HVA-001
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: G.Senti, University of Zurich
Other Study IDs: ZU-HVA-001
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2008-09

CONDITIONS: Hymenoptera Sting Allergy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Hymenoptera sting allergic patients under immunotherapy
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of sting frequency

SUMMARY:
In Switzerland, 3.5% of the population are suffering from hymenoptera venom allergy. The only causal treatment of hymenoptera alelrty is venom specific immunotherapy. There are however several reasons, which question the relatively broad application of this expensive treatment. That's why we aim at investigating the actual risk for hymenoptera stings in patients undergoing allergen specific immunotherapy against hymenoptera sting allergy

ELIGIBILITY:
Inclusion criteria:

* Bee and/or Wasp allergic patients treated by SIT

Exclusion criteria:

* None

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hymenoptera sting allergic patients under allergen specific immunotherapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland